CLINICAL TRIAL: NCT05402709
Title: Comparison of the Effectiveness of Posterior Capsule Stretching and Posterior Mobilization on Subacromial Impingement Syndrome
Brief Title: Effectiveness of Posterior Capsule Stretching and Posterior Mobilization on Subacromial Impingement Syndrome
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Yeditepe University (Other)
Responsible Party: Principal Investigator, Ebru Akbuğa Koç, Principal investigator, Yeditepe University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2016-11/03
Record Dates: First submitted 2022-05-28; First posted 2022-06-02 (Actual); Last update posted 2022-11-08 (Actual); Status verified 2022-11

CONDITIONS: Subacromial Impingement Syndrome
Keywords: subacromial impingement syndrome; posterior capsule; mobilisation
MeSH Terms: conditions — Shoulder Impingement Syndrome

STUDY DESIGN:
Intervention Model Description: Individuals were randomly divided into 3 different groups as posterior mobilisation, posterior capsule stretching and control group
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Posterior mobilization group (Active Comparator): Posterior mobilization, classical stretching, strengthening exercises were applied and home exercise program were given
  Interventions: Other: Posterior mobilisation technique
- Posterior capsule stretching (Active Comparator): Posterior capsule stretching, classical stretching, strengthening exercises were applied and home exercise program were given
  Interventions: Other: Posterior capsule stretching
- Control group (No Intervention): No treatment was given, only assessment of posterior capsule tightness was applied.

INTERVENTIONS:
Other: Posterior mobilisation technique — Posterior mobilisation technique were applied
  Arms: Posterior mobilization group
Other: Posterior capsule stretching — Posterior capsule stretching were applied
  Arms: Posterior capsule stretching

SUMMARY:
Subacromial Impingement Syndrome is one of the most common shoulder pathologies causing shoulder pain, functional disability and reduced quality of life. This study was designed to investigate the effectiveness of posterior capsule stretching and posterior mobilization on shoulder joint functions in Subacromial Impingement Syndrome.

DETAILED DESCRIPTION:
Subacromial Impingement Syndrome is one of the most common shoulder pathologies causing shoulder pain, functional disability, and reduced quality of life. This study investigated the effectiveness of posterior capsule stretching and posterior mobilization on shoulder joint functions in Subacromial Impingement Syndrome.

74 patients with SIS were enrolled, 58 were included, but 50 completed the study. Also, 30 healthy individuals were included and completed the study. The introductory characteristics of cases with the sociodemographic survey, pain intensity with VAS, upper extremity function with American Shoulder and Elbow Surgeons Standardized Shoulder Assessment Form and Modified Constant Murley Score, upper extremity disability and health situation with Quick Disability Arm, Shoulder and Hand Score, the evaluation of musculoskeletal symptoms with Cornell Musculoskeletal Discomfort Questionnaire, range of motion with a goniometer, shoulder muscle strength with myometer, grip strength with dynamometer and pinch meter and posterior capsule tightness with a tapeline. Individuals were divided into three different groups posterior mobilisation, posterior capsule, and control group. While participants included in the mobilization group were given classical stretching and strengthening and home exercise programs in addition to posterior mobilization, for the capsule stretching group, classical stretching and strengthening and home exercise program were given in addition to posterior capsule stretching exercise, and no exercise program was given to the control group and only posterior capsule tightness evaluation was applied.

In this study, while there was found a statistically significant difference between both groups in the Constant score and involved part External Rotation range of motion (p<0,05), a statistically significant difference was not observed in the evaluation of muscle strength, grip strength and posterior capsule tightness (p>0,05). In the participants who applied mobilization, the functional capacity of the shoulder joint was increased more than those of the capsule stretching.

ELIGIBILITY:
Inclusion Criteria:

* To be between 30-60 years old
* Positive Neer, Hawkins-Kennedy impingement tests
* Painful arch and minimal limitation during active flexion and abduction movements in the glenohumeral joint area or proximal arm
* Symptoms lasting longer than 1 month

Exclusion Criteria:

* Adhesive capsulitis,
* Rotator cuff tears,
* Calcific tendinitis findings in radiology,
* Having a heart disease
* Presence of neurological diseases,
* Cognitive and mental problems that will affect understanding,
* Cervical radiculopathies,
* Presence of inflammatory joint diseases,
* Surgical intervention on the same shoulder in the last 12 months,
* To have had physical therapy on the same shoulder in the last 3 months,
* Presence of instability or previous dislocation history.

Ages: 30 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 80 (Actual)
Dates: Start 2016-12-26 (Actual); Primary Completion 2017-02-08 (Actual); Study Completion 2017-06-25 (Actual)

PRIMARY OUTCOMES:
Assessment of Joint Range of Motion | 6 weeks
  Shoulder flexion, abduction, external and internal rotations were evaluated actively and passively using a classical goniometer (Santa Pharma 12 inch) while the patient was in the supine position. Measurements were made twice, before and at the end of the treatment (6th week), and the average value was taken bilaterally three times.
Assessment of Muscle Strength | 6 weeks
  "JTech Commander Power Track IITM" Myometer device was used for muscle strength evaluation. In the evaluation, shoulder flexion, extension, abduction, internal and external rotation movements were held with resistance for 3-5 seconds for each movement (according to the manual muscle test rules). Measurements were made twice, before and after the treatment. Each measurement was repeated bilaterally and three times, and the average values were taken and tested by the physiotherapist.
Assessment of Grip Strength | 6 weeks
  The grip strength of the hand was evaluated using the "JTech Commander Grip Track Hand Dynamometer". The patient was evaluated by the physiotherapist in a sitting position in a chair, with the shoulder to be tested in adduction and neutral rotation, the elbow in 90 degree flexion, and the forearm and wrist in neutral position. The patients were asked to squeeze the dynamometer as hard as possible. After a 30-second rest break between measurements, the next measurement was started. Measurements were made twice, before and after the treatment. Each measurement was repeated bilaterally and three times and evaluated by taking the average values.
Assessment of Pain | 6 weeks
  The pain intensity of the patients was evaluated with the Visual Analogue Scale (VAS) by the physiotherapist. The Visual Analogue Scale is a scale in which evaluation is made on a 10 cm line drawn on the horizontal plane with a maximum of 10 and a minimum of 0 points. The patient was asked to mark the severity of the pain he felt in his shoulder on this line, and the pain before and after the treatment was evaluated with this method.
American Shoulder and Elbow Surgeons Assessment Form | 6 weeks
  The American Shoulder and Elbow Surgeons Assessment Form (ASES) is a standard shoulder evaluation form that evaluates pain and function in the upper extremity, including objective and subjective parts, prepared by shoulder and elbow surgeons. The questionnaire consists of pain (VAS) and function (10 questions). The function section consists of a 4-point Likert scale for each question. The Turkish version of ASES was used in the study, the validity and reliability of which were made by Çelik et al. in 2012. The total score of the questionnaire completed by the patients before and after the treatment was evaluated out of 100.
Quick-DASH | 6 weeks
  The Arm, Shoulder and Hand Problems Questionnaire (Quick-DASH) is a scale that evaluates the disability and health status of the upper extremity, which can be filled by the individual alone. The questionnaire consists of 11 questions, each of which evaluates problems such as whether the patient has limitations in activities that require upper extremity functions in daily life activities, the effect of the current problem on the person's social activities, pain, tingling sensation and difficulty in sleeping, and a business model with 4 questions each, and sports that require high performance. The questions do not only address the shoulder area, but also cover the hand and arm. Scoring takes a value between 0-100 and a high score reflects more disability. In our study, we made use of the website while performing the Quick-DASH scoring. People with Subacromial Impingement Syndrome completed this questionnaire at the beginning and end of treatment.
Modified Constant-Murley Score (CMS) | 6 weeks
  Constant Murley Score (CMS), the first shoulder scoring system developed, was put into effect in 1987 by Constant and Murley. This questionnaire, which is used to evaluate various diseases of the shoulder; pain, activities of daily living, strength and range of motion are evaluated qualitatively and quantitatively. The CMS consists of pain (15 points), activities of daily living (20 points), movement (40 points), and strength (25 points) subscales. The difference of the modified CMS from the original CMS; While the VAS was used for the pain scale in the modified CMS, the pain was rated as "severe", "moderate", "mild", and "absent" in the original. Modified CMS is scored over 100 points. A higher score indicates higher quality of functionality. We also used the Turkish version of Modified Constant-Murley Score at the beginning and end of the treatment in our study.
Cornell Musculoskeletal Discomfort Questionnaire | 6 weeks
  The Cornell Musculoskeletal Discomfort Questionnaire is a data collection tool developed at the Human Factors and Ergonomics Laboratory at Cornell University and used to evaluate musculoskeletal problems. The Cornell Musculoskeletal Disorders Questionnaire includes questions such as the frequency and severity of musculoskeletal disorders and whether these disorders interfere with work, over 10 upper extremity body regions on 3 separated scales. In our study, the Turkish version of the Cornell Musculoskeletal Discomfort Questionnaire was used, and it was filled in by the patients at the beginning and end of the treatment.
Assessment of Posterior Capsule Tightness | 6 weeks
  The medial epicondyle of the tested arm is marked with a pencil and aligned with the subject's acromion perpendicular to the treatment table with the spine in a neutral position. By stabilizing the lateral border of the scapula while the shoulder is in the retracted position, scapular movement is restricted and the subject's humerus is positioned at 90° horizontal abduction, 0° rotation at the start of the test.